CLINICAL TRIAL: NCT01362426
Title: A Quality Use of Medicine Clinical Registry to Assess Clinical Outcomes in Patients With Schizophrenia Treated With Intramuscular Injections of Paliperidone Palmitate
Brief Title: Paliperidone Palmitate Effectiveness Assessment Registry - Longitudinal (PEARL)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR018013
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; paliperidone palmitate; INVEGA SUSTENNA; registries; quality of healthcare
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: paliperidone palmitate Dosage and administration will be according to the paliperidone palmitate approved Australian Product Information.
  Interventions: Drug: paliperidone palmitate

INTERVENTIONS:
Drug: paliperidone palmitate — Dosage and administration will be according to the paliperidone palmitate approved Australian Product Information.

SUMMARY:
The primary objective of this study is to determine if Australian patients with schizophrenia treated with paliperidone palmitate under conditions of continuous monitoring of outcomes over a 12-month period achieve relapse rates comparable to published literature.

DETAILED DESCRIPTION:
This study involves the establishment of PEARL, an Australian Quality Use of Medicine clinical registry designed to collect clinical and social data on up to 300 patients with schizophrenia for a 12-month period after initiating treatment with intramuscular (IM) injections of paliperidone palmitate as part of their routine clinical care. Continuous feedback of clinical outcomes will be via regular reports to all registry sites. Enrollment in PEARL should be considered only after the clinical decision to prescribe IM paliperidone palmitate has already been made because the treating physician has determined that this treatment is the best option for the patient. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Must fulfill the diagnostic criteria for Schizophrenia Disorders as defined by Diagnostic and Statistical Manual of Mental Disorders Version IV (DSM-IV)
* Must meet the approved Therapeutic Goods Administration (TGA) indication for injectable paliperidone palmitate
* Must have provided written informed consent indicating that they understand the purpose of and procedures required for the registry and are willing to participate in the registry.

Exclusion Criteria:

* Those with a known hypersensitivity to either paliperidone or risperidone, or to any excipients in the paliperidone palmitate formulation
* Employees of the clinician or study centre, with direct involvement in the proposed registry or other studies under the direction of that clinician or study centre, as well as family members of the employees or the clinician.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Australian patients with schizophrenia will be enrolled in the registry
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with symptomatic relapse | Up to 12 months

SECONDARY OUTCOMES:
Clinical effectiveness and social outcomes as measured by the following clinical assessment tools: CGI-S. | Up to 12 months
Clinical effectiveness and social outcomes as measured by HoNOS. | Up to 12 months
Clinical effectiveness and social outcomes as measured by PSP. | Up to 12 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 12 months
Clinical effectiveness and social outcomes as measured by the following clinical assessment tools: GAF | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd
Locations (10):
- Australia (10):
  - Bendigo
  - Box Hill
  - Elizabeth Vale
  - Epping
  - Fitzroy
  - Fremantle
  - Glenside
  - Meadowbrook
  - Waratah
  - Wollongong